CLINICAL TRIAL: NCT07176260
Title: Diagnostic and Prognostic Significance of Circulating Oxidative Stress and Blood Cell Mitochondrial Respiration in Pre-Capillary Pulmonary Hypertension
Brief Title: Exploring Blood Cell Function and Oxidative Stress to Improve Diagnosis and Treatment in Pre-Capillary Pulmonary Hypertension
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: CE 2017-24
Record Dates: First submitted 2025-09-08; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Pre-capillary Pulmonary Hypertension
Keywords: Mitochondrial respiration; Oxidative stress; PBMCs, platelets; Pulmonary arterial hypertension; Pulmonary hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * Whole blood - collected from peripheral veins or from jugular vein during right heart catheterization.
  * Plasma/serum - separated from blood samples for biochemical and oxidative stress analyses.
  * White blood cells (PBMCs) - isolated from whole blood for mitochondrial respiration studies and related assays.
  * Platelets - isolated from whole blood for mitochondrial respiration studies and related assays.
  * Arterialized and arterial blood - obtained from the pulmonary artery occlusion site during catheterization for comparative mitochondrial and oxidative stress analyses
  No other biospecimens (e.g., urine, tissue) will be collected or retained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patients with pre-Capillary pulmonary hypertension — Patients will be followed for 3 years with routine clinical, hemodynamic, and laboratory assessments. Blood samples for oxidative stress and mitochondrial function analyses will be collected during scheduled follow-up visits or catheterization procedures. No intervention beyond standard care will be performed.

SUMMARY:
This study aims to understand how blood cell (including peripheral blood mononuclear cells ((PBMCs) or platelets) function and oxidative stress can help physicians detect and predict the course of pre-capillary pulmonary hypertension. We hypothesize that changes in the mitochondrial function of blood cells and oxidative stress may be early markers of disease progression and severity.

The study will also explore how these blood markers relate to routine clinical and heart function measurements, such as echocardiography, right heart catheterization, 6-minute walk tests, and functional status, to see if they can help monitor patients over time and guide personalized care.

This is a non-interventional study. Blood samples will be collected during routine visits planned for diagnosis and follow-up. The study will include 120 patients diagnosed with pre-capillary pulmonary hypertension, who will be followed for 3 years. Blood samples will be taken up to three times per year to measure mainly oxidative stress and mitochondrial function in blood cells. These measurements will be compared with clinical tests to see if they can help predict the course of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) diagnosed with pre-capillary pulmonary hypertension confirmed by right heart catheterization
* Patients classified according to the international clinical classification:

  * Group 1: Pulmonary arterial hypertension (PAH)
  * Group 3: Pulmonary hypertension associated with chronic respiratory diseases and/or hypoxia
  * Group 4: Chronic thromboembolic pulmonary hypertension (CTEPH)
* Patients scheduled for routine clinical follow-up and/or right heart catheterization at the study center.
* Ability and willingness to provide informed consent for participation and data analysis.

Exclusion Criteria:

* Postcapillary pulmonary hypertension (pulmonary arterial wedge pressure >15 mmHg).
* Conditions precluding safe blood sampling (e.g., severe anemia, coagulopathy).
* Patients already enrolled in interventional clinical trials that could interfere with mitochondrial or oxidative stress measurements
* Patients unable or unwilling to provide informed consent
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prevalent or incident patients with pre-capillary pulmonary hypertension
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Blood Cell Mitochondrial Function and Respiration and Oxidative Stress Markers | 3 years
  Analyse Blood Cell Mitochondrial Function and Respiration and Oxidative Stress Markers

SECONDARY OUTCOMES:
Correlation of blood cell mitochondrial function and respirations and oxidative stress markers | 3 years
  Correlation of blood cell mitochondrial function and respirations and oxidative stress markers with routine clinical and hemodynamic parameters, including echocardiography, right heart catheterization, 6-minute walk test (6MWT), NYHA functional class, and BNP or NT-pro BNP levels

CONTACTS AND LOCATIONS:
Overall Officials: Marianne RIOU, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Hôpitaux Universitaires de Strasbourg - Service Physiologie explorations fonctionnelles, Strasbourg, Bas-Rhin, France

IPD SHARING:
Plan to Share IPD: Undecided